CLINICAL TRIAL: NCT01574430
Title: A Randomized, Double-masked, Multicenter, Controlled Study of Photodynamic Therapy in Patients With Central Serous Chorioretinopathy
Brief Title: Study of Photodynamic Therapy (PDT) in Patients With Central Serous Chorioretinopathy (CSC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Mingwei Zhao, Dr., Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDTCSC-CHINA
Record Dates: First submitted 2012-04-08; First posted 2012-04-10 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — 1-phenyl-3,3-dimethyltriazene; Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50% dose PDT (Active Comparator): patients in this group was given 50% verteporfin dose PDT
  Interventions: Procedure: PDT
- 30% dose PDT (Experimental): patients in this group was given 30% verteporfin dose PDT
  Interventions: Procedure: PDT

INTERVENTIONS:
Procedure: PDT — 30% or 50% verteporfin dose PDT was given to patients with CSC
  Other Names: photodynamic therapy

SUMMARY:
The purpose of this study is to determine the safety and efficacy of PDT at 30% verteporfin dose in the treatment of CSC.

ELIGIBILITY:
Inclusion Criteria:

* patients with CSC
* patients signed the ICF
* patients with course of CSC less than 6 months
* patients did not undertake any treatment for CSC

Exclusion Criteria:

* patients with porphyria
* patients allergic to verteporfin
* pregnant or nursing women
* poor patients compliance
* sever liver dysfunction
* dioptric media opacities which make it difficult to exam fundus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BCVA | 1 week,2 weeks,3 weeks,1 month,3months, 6 months, 1 year

SECONDARY OUTCOMES:
Leakage at RPE level in FA | 1 week
Change from baseline in central retinal thickness | 1 week,2 weeks,3 weeks,1 month,3months, 6 months, 1 year
The incidence rate of adverse event | 1 week,2 weeks,3 weeks,1 month,3months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei Zhao, M.D, Study Director — Peking University People's Hospital; Youxin Chen, M.D, Principal Investigator — Peking Union Medical College; Feng Zhang, M.D, Principal Investigator — Beijing Tongren Hospital of Capital Medical University; Hong Dai, M.D, Principal Investigator — Beijing Hospital; Xiaoxin Li, M.D, Study Chair — Peking University People's Hospital
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203
- [Derived] Zhao M, Zhang F, Chen Y, Dai H, Qu J, Dong C, Kang X, Liu Y, Yang L, Li Y, Zhou P, Pan CT, Zhang L, Liu P, Zhou H, Jiao X, Xiong Y, Tian R, Lu Y, Yu X, Li X. A 50% vs 30% dose of verteporfin (photodynamic therapy) for acute central serous chorioretinopathy: one-year results of a randomized clinical trial. JAMA Ophthalmol. 2015 Mar;133(3):333-40. doi: 10.1001/jamaophthalmol.2014.5312. PMID 25555191